CLINICAL TRIAL: NCT01933854
Title: ASSESSMENT OF URINARY INCONTINENCE IN WOMEN AT AMAPA STATE: COMPARISON BETWEEN URBAN AND RIVERSIDE POPULATIONS
Brief Title: Urinary Incontinence in Women From Amapa
Acronym: iuemcp
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Jorge Milhem Haddad, Phd, University of Sao Paulo General Hospital
Other Study IDs: 2012MACAPASP
Record Dates: First submitted 2013-06-18; First posted 2013-09-02 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Urinary Incontinence
Keywords: Urinary incontinence; riverside; women; Amapa
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: None Retained — Urban group: women aged 20 years or over, who are not pregnant and are looking for a health facility to perform womb cancer prevention exam in Macapa, the capital city of the Amapa State.
  Riverside Group: Women aged 20 years or over, who are not pregnant and are looking for a health facility to perform womb cancer prevention exam on the Bailique Island.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Riverside group: Women aged 20 years or over who are not pregnant living riverside area of the Amapa State Brazil.
- urban group: women aged 20years or over not pregnant and living urban area

SUMMARY:
The investigators aim to study the prevalence of urinary incontinence in women who live in the riverside community in the state of Amapa (The Bailique Island) and compare it to the prevalence of urinary incontinence in women who live in the urban region -Macapa-the capital city of the Amapa State - Brazil.

DETAILED DESCRIPTION:
The study aims to compare urinary complaints of women belonging to two different groups: women who live in a riverside area of the Amapa State-the Bailique Island, which is about 12 hours by boat from the state capital city and compare them to those of the women who live in the urban region -Macapa (the capital city of the Amapa State). The main goals are: to describe the clinical features of the women in the study, assess probable risk factors concerning the urinary incontinence, make physical gynecological exam as well as urodynamic studies in the patients who have urinary complaints and use a life quality questionnaire with those patients (Kings Health Questionnaire).

Cross and prevalence Study, followed by case series. Cohort study between the two populations. The riverside group with 120 interviews and the urban group with 260 interviews, where the sample calculation was based on the population of each region and the incidence of urinary incontinence checked through a pilot study.

After reading and signing an informed consent, interviews with women aged 20 years or over and non-pregnant are hold so as to identify those who have complaints about urinary incontinence, socio-economic data and risk factors. In patients who complain about urinary incontinence, gynecological exams are performed in order to assess genital prolapse and urodynamic studies are made as to confirm urinary incontinence and life quality questionnaire. All the data will be encoded in the database and analyzed through statistics programs and a comparison between the two groups (urban and riverside) will be made.

ELIGIBILITY:
Inclusion Criteria:

* women aged 20 or over
* living either in the urban area or in the riverside

Exclusion Criteria:

* women under 20 and
* pregnant

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Urban group: women aged 20 years or over, who are not pregnant and are looking for a health facility to perform womb cancer prevention exam in Macapa, the capital city of the Amapa State.
  Riverside Group: Women aged 20 years or over, who are not pregnant and are looking for a health facility to perform womb cancer prevention exam on the Bailique Island.
Sampling Method: Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-09 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Urinary incontinence and life style (riverside population X urban population) | Thirteen months
  Assessment of urinary incontinence in women who live in a riverside community and who have had a home dilivery when compared with women from urban community. They will be assessed through the use of a questionnaire of quality of life and urodynamic evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Aljerry Rego, Graduate, Principal Investigator — University of Sao Paulo
Locations (1):
- Mae Luzia Women's Hospital, Macapá, Amapá, Brazil